CLINICAL TRIAL: NCT04202120
Title: Age Stereotype Priming and Moderating Effects of Social Participation
Brief Title: Age Stereotype Priming and Social Participation
Acronym: ASPSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AFC2018
Record Dates: First submitted 2019-12-15; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Aging Well; Memory Loss
Keywords: Age stereotypes; episodic memory; social participation
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Age-related priming (Experimental): Participants received a review of the profile of their social participation. They also received psycho-education about memory components. They were give given memory tests with age-related primes.
  Interventions: Other: Age-related stereotyping priming
- Non-age related priming (Active Comparator): Participants received a review of the profile of their social participation. They also received psycho-education about memory components. They were give given memory tests with NON age-related primes.
  Interventions: Other: Non age-related stereotype priming

INTERVENTIONS:
Other: Age-related stereotyping priming — The priming intervention was performed using the E-prime 2.0 software (Psychology Software Tools, Pittsburgh, PA). To ensure the primes flashed on screen were beyond awareness, the similar adjustment procedure was taken (see Levy, 1996; Stein et al., 2002). After the trial block, participants were asked to try to report any words viewed during each trial. The stimulus onset asynchrony (SOA) will be reduced or enhanced whenever 2 words or above were correctly reported or no single word could be reported respectively. The priming SOA for this study ranged from 32 ms to 208 ms (M = 98.70 ms. SD = 48.60).
  Arms: Age-related priming
Other: Non age-related stereotype priming — he priming intervention was performed using the E-prime 2.0 software (Psychology Software Tools, Pittsburgh, PA). To ensure the primes flashed on screen were beyond awareness, the similar adjustment procedure was taken (see Levy, 1996; Stein et al., 2002). After the trial block, participants were asked to try to report any words viewed during each trial. The stimulus onset asynchrony (SOA) will be reduced or enhanced whenever 2 words or above were correctly reported or no single word could be reported respectively. The priming SOA for this study ranged from 32 ms to 208 ms (M = 98.70 ms. SD = 48.60).
  Arms: Non-age related priming

SUMMARY:
Memory performance is shown to be affected by age stereotypes among older adults. The purpose of the study is to examine the effects of age stereotype primes on episodic memory using priming intervention. The moderating effects of social participation is also examined.

DETAILED DESCRIPTION:
All participants are community-dwelling older adults residing in Hong Kong. They are invited to review their social participation profile and given a brief psycho-education about memory.

They are then randomly allocated to one of the two following conditions. Participants are primed either with age stereotypes or non-age stereotypes words by implicit priming intervention in the context of a reaction task prior to the episodic memory tasks. Other measures such as demographic variables and social participation rate are collected by questionnaire during the delayed recall interval.

ELIGIBILITY:
Inclusion Criteria:

Indication of largely normal cognitive functioning as screened on the Montreal Cognitive Assessment (MoCA) with Hong Kong norms -

Exclusion Criteria:

Sensory deficits and evidence of cognitive impairment as screened on the Montreal Cognitive Assessment (MoCA) with Hong Kong norms

-

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-01-12 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Hong Kong List Learning Test | Change from baseline through study completion, an average of 2 hours
  The Hong Kong List Learning is a validated tool for assessing episodic memory for aged Chinese speaking adults (Chan, 2006). It was further taken for investigating differences among older adults with normal cognitive ability and older adults with mild cognitive impairment (Yeung et al., 2016). The random control list was taken in this study. It comprises 16 words formed by four categories:

CONTACTS AND LOCATIONS:
Overall Officials: Alma Au, PhD, Study Chair — Dr (female)
Locations (1):
- Applied Social Sciences, Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Au A, Chan AS, Chiu H. Verbal learning in Alzheimer's dementia. J Int Neuropsychol Soc. 2003 Mar;9(3):363-75. doi: 10.1017/S1355617703930025. PMID 12666761
- [Background] Wong A, Yiu S, Nasreddine Z, Leung KT, Lau A, Soo YOY, Wong LK, Mok V. Validity and reliability of two alternate versions of the Montreal Cognitive Assessment (Hong Kong version) for screening of Mild Neurocognitive Disorder. PLoS One. 2018 May 23;13(5):e0196344. doi: 10.1371/journal.pone.0196344. eCollection 2018. PMID 29791452
- [Background] Stein R, Blanchard-Fields F, Hertzog C. The effects of age-stereotype priming on the memory performance of older adults. Exp Aging Res. 2002 Apr-Jun;28(2):169-81. doi: 10.1080/03610730252800184. PMID 11928527
- [Derived] Chan SCY, Au AML, Lai SMK. The detrimental impacts of negative age stereotypes on the episodic memory of older adults: does social participation moderate the effects? BMC Geriatr. 2020 Nov 5;20(1):452. doi: 10.1186/s12877-020-01833-z. PMID 33153433